CLINICAL TRIAL: NCT00129012
Title: Self-Gated Breath-Hold Technique for Helical Tomotherapy in Patients With Non-Small Cell Lung Cancer: A Feasibility Study
Brief Title: Self-Gated Breath-Hold Technique for Helical Tomotherapy in Patients With Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LU-11-0051 / 21808
Record Dates: First submitted 2005-08-09; First posted 2005-08-11 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2012-03

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: radiation therapy; carcinoma; non-small cell lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Tomotherapy

SUMMARY:
Non-small cell lung cancer (NSCLC) is a disease that often cannot be surgically operated on. As a result, treating the tumor with radiation has become the main standard of treatment. Radiation therapy though, is limited by various factors, including the difficulty in properly imaging the lung tumor since the lung can move up to 4 cm between breathing in and out. Consequently, a radiation oncologist must consider a larger area of the lung to treat with radiation - increasing the amount of normal tissue exposed to harmful rays and therefore leading to increased side-effects. Two techniques being explored into improving tumor management while minimizing the side effects in NSCLC are breath-held gating and tomotherapy. Breath-held gating is a technique for consistently imaging the tumor at the right moment in a patient's breathing cycle - decreasing the normal tissue exposed to harmful radiation. Tomotherapy, a new technique in delivering radiation, will further allow the investigators to focus treatment on the tumor and exclude more normal tissues. Therefore, they hope that these methods will prove to be a better way in treating people with NSCLC.

DETAILED DESCRIPTION:
Non-small cell lung cancer (NSCLC) is a disease that often presents as an unresectable tumor. As a result, radiotherapy is the main standard of treatment. Unfortunately, radiotherapy is limited by several factors, including that the lung can move up to 4 cm between inspiration and expiration. As a result, a radiation oncologist often has to widen his treatment field to include for this motion. This leads to greater side effects for the patient. Two techniques that are being explored to improve the tumor control of radiotherapy and to minimize side effects to normal tissues in NSCLC treatment include breath-held gating and tomotherapy. Breath-held gating will allow the investigators to treat patients at the right moment in their breathing cycle consistently - minimizing the normal tissue exposed to radiation. In addition, both gated breathing and tomotherapy will allow the investigators to create a more refined tumor volume treated and exclude more of the normal tissues. Consequently, they hope these methods will prove to be a better way to treat patients with non-resectable NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Stage I-III NSCLC
* Karnofsky Performance Status (KPS) equal to or greater than 70
* Forced expiratory volume in 1 second (FEV1) equal to or greater than 1.0L

Exclusion Criteria:

* Myocardial infarction (MI) disease
* Recurrent disease
* Complete tumour resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-04; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
safety and adverse events

SECONDARY OUTCOMES:
efficacy and survival

CONTACTS AND LOCATIONS:
Overall Officials: Wilson Roa, MD, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada